CLINICAL TRIAL: NCT06851676
Title: Functional and Metabolic Effects of Fonte Fausta® Water on the Musculoskeletal System in Patients with Osteoporosis/Osteopenia with or Without Sarcopenia
Brief Title: Functional and Metabolic Effects of Fonte Fausta® Water on Bone and Muscle Health in Osteoporotic Patients
Acronym: FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANTIMO (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor-Investigator, ANTIMO, professor, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOCUS01
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-07

CONDITIONS: Osteopenia, Osteoporosis; Sarcopenia
Keywords: osteoporosis; sarcopenia; functioning; calcium; water
MeSH Terms: conditions — Bone Diseases, Metabolic; Sarcopenia; Osteoporosis | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): Enrolled patients will be divided into three groups: patients with osteoporosis/osteopenia accompanied by sarcopenia, patients with osteoporosis/osteopenia without sarcopenia, and a control group with non-osteometabolic conditions. Each group has been randomized into two subgroups: one receiving Fonte Fausta® and the other receiving natural mineral water.
  Interventions: Dietary Supplement: water supplemented by calcium
- control (Placebo Comparator): Enrolled patients will be divided into three groups: patients with osteoporosis/osteopenia accompanied by sarcopenia, patients with osteoporosis/osteopenia without sarcopenia, and a control group with non-osteometabolic conditions. Each group has been randomized into two subgroups: one receiving Fonte Fausta® and the other receiving natural mineral water.
  Interventions: Other: Water (Placebo)

INTERVENTIONS:
Dietary Supplement: water supplemented by calcium — Fonte Fausta® water is a natural mineral water, rich in essential minerals, such as calcium, magnesium, and bicarbonate, which are important for maintaining bone density, muscle function, and overall metabolic health.
  Arms: intervention
Other: Water (Placebo) — a natural mineral commercially available
  Arms: control

SUMMARY:
This clinical study investigates the effects of Fonte Fausta® water on bone and muscle metabolism, as well as quality of life, in patients with osteoporosis or osteopenia, with or without sarcopenia. Conducted as a multicenter, triple-arm trial, it evaluates functional and biochemical markers over 12 months. Patients are randomized into groups receiving either Fonte Fausta® or standard mineral water, with assessments including laboratory tests, bioimpedance analysis, physical and nutritional evaluations, bone density measurements, and quality of life surveys.

DETAILED DESCRIPTION:
This study aims to determine the impact of Fonte Fausta® water on bone and muscle metabolism in patients with osteoporosis or osteopenia, with or without sarcopenia, over a 12-month period. The research follows ethical guidelines (Helsinki Declaration) and has been approved by the Ethics Committee of the University of Campania "Luigi Vanvitelli." All participants provided informed consent.

Study Design and Participants The study is a multicenter, triple-arm interventional clinical trial conducted at the University of Campania "Luigi Vanvitelli." Participants include individuals diagnosed with primary osteoporosis or osteopenia, with or without sarcopenia, based on clinical guidelines and the EWGSOP2 criteria. Osteoporosis is diagnosed by a BMD T-score ≤ -2.5 SD or the presence of a fragility fracture, while osteopenia is defined as a BMD T-score between -1 and -2.5 SD. Sarcopenia diagnosis is based on low muscle strength and low muscle mass.

Exclusion criteria include secondary osteoporosis causes (e.g., chronic diseases, endocrine disorders, long-term corticosteroid use), psychiatric conditions affecting consent, and pregnancy or breastfeeding.

Study Groups and Randomization

Participants are divided into three primary groups:

Patients with osteoporosis/osteopenia and sarcopenia Patients with osteoporosis/osteopenia without sarcopenia A control group with non-osteometabolic conditions

Each group is further randomized into two subgroups:

One receiving Fonte Fausta® water One receiving natural mineral water Assessments and Evaluations

Participants undergo evaluations at three time points:

Baseline (T0) Six months (T6) Twelve months (T12)

Key assessments include:

Laboratory Tests: Blood and urine analyses to assess biochemical markers such as ALP, bone-specific ALP, PTH, 25(OH)D3, and CTX.

Bioimpedance Analysis (BIA): Measures body composition, including fat and muscle mass.

Physical and Nutritional Assessments: Includes questionnaires like the International Physical Activity Questionnaire, handgrip strength measurements, and the Mini Nutritional Assessment.

Bone Health and Fall Risk: DXA scans measure BMD, and the FRAX® algorithm estimates fracture risk.

Pain, Performance, and Quality of Life: Evaluations include the Short Physical Performance Battery (SPPB), Brief Pain Inventory (BPI), and quality of life questionnaires (EQ-5D-3L and EQ-VAS).

This study aims to determine whether Fonte Fausta® water offers functional and metabolic benefits for bone and muscle health, potentially improving quality of life and reducing fracture risk in osteoporotic and osteopenic patients.

ELIGIBILITY:
Inclusion Criteria:

-a diagnosis of primary osteopenia or osteoporosis , with or without sarcopenia, based on the latest clinical practice guidelines and EWGSOP2 criteria .

Exclusion Criteria:

* secondary causes of osteoporosis (such as prolonged high-dose glucocorticoid use, liver or kidney disease, cancer, neurodegenerative or inflammatory diseases, chronic obstructive pulmonary disease, and endocrine disorders)
* psychiatric disorders that could impair informed consent
* pregnancy or breastfeeding.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Bioimpedance Analysis (BIA) | 0 (T0), 180 (T1), and 365 days (T2)
  Bioimpedance Analysis (BIA) is a non-invasive method used to assess body composition, including fat mass, muscle mass, and total body water. It works by measuring the resistance of electrical currents as they pass through the body's tissues, with lean tissues (muscle and water) conducting electricity better than fat tissues.

SECONDARY OUTCOMES:
Laboratory Tests | 0 (T0), 180 (T1), and 365 days (T2)
  Blood samples (20 ml), a 24-hour urine collection, and early morning urine analyses will be conducted to evaluate key biochemical markers, including ALP, bone-specific ALP, PTH, 25(OH)D3, CTX, among others.

CONTACTS AND LOCATIONS:
Locations (1):
- Vico de Crecchio, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
data will be shared upon reasonable request
Supporting Information: Study Protocol